CLINICAL TRIAL: NCT05344300
Title: Temperature Recording in Lungs of Volunteers With and Without Pulmonary Diseases
Acronym: TEMP-REC-LUNG
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chronic Obstructive Pulmonary Disease Trial Network, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: TEMP-REC-LUNG
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Temperature Change, Body; Bronchiectasis; Heat Exposure; Heat
MeSH Terms: conditions — Body Temperature Changes; Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lung-healthy group
  Interventions: Other: Temperature-measurement in lungs under sauna bath
- Bronchiectasis group
  Interventions: Other: Temperature-measurement in lungs under sauna bath

INTERVENTIONS:
Other: Temperature-measurement in lungs under sauna bath — Through a bronchoscopy procedure under an 88-92℃ environment, the air temperature is measured in the 1st, 2nd and 3rd bronchial segment, at 4th and 5th bronchial segment and at 6th-10th bronchial segment in resp. the right and left lung. The temperature is measured at time: 0 seconds (s), 15 s, 30 s, 45 s, 60 s, 75 s, 90 s, 105 s, 120 s, 135 s and 150 s.

SUMMARY:
The purpose of the project is to estimate the air temperature in the lungs after a change from room temperature (25℃) to an environment with a constant temperature of 88-92℃ in resp. lung-healthy persons and persons with bronchiectasis.

DETAILED DESCRIPTION:
Heat is a widely available therapeutic modality and is often used for recovery after physical activity and pain treatment, and sauna bathing is a form of whole body thermotherapy ranging from 80-100 ℃ and low humidity of 10-20%. The heat load in a sauna has been shown to activate several beneficial physiological effects, and no adverse effects on the lungs have been demonstrated. It is unknown how much the air temperature in the lower respiratory tract (bronchial tree) in humans rises to under surroundings of 88-92℃.

This is an observational, clinical trial investigating the changes in air temperature at different bronchial segments in both lungs under surroundings of 88-92℃ resp. in lung-healthy persons and persons with bronchiectasis.

ELIGIBILITY:
Lung-healthy group:

Inclusion criteria:

* Age ≥ 18 years
* Competent and capable
* Forced expiratory volume in the first second (FEV1)>1,0 L
* Does not suffer from bronchiectasis, asthma, chronic obstructive pulmonary disease, pulmonary fibrosis, sarcoidosis, active lung infection (past 30 days) or lung cancer

Exclusion criteria:

* Allergy to lidocaine and/or midazolam
* Contraindications to bronchoscopy*
* Previous severe laryngospasm (intubation requiring)
* Pregnancy/breastfeeding
* Severe linguistic problems or inability to give informed consent
* Severe mental illness that is not controlled with medication. NB: Patients with controlled mental illness can be included and will be asked on an equal footing as others

Bronchiectasis group:

Inclusion criteria:

* Age ≥ 18 years
* Competent and capable
* FEV1>1,0 L
* Have diagnosed bronchiectasis [radiology verified and evaluated by pulmonary specialist]

Exclusion criteria:

* Allergy to lidocaine and/or midazolam
* Contraindications to bronchoscopy*
* Previous severe laryngospasm (intubation requiring)
* Pregnancy/breastfeeding
* Severe linguistic problems or inability to give informed consent
* Severe mental illness that is not controlled with medication. NB: Patients with controlled mental illness can be included and will be asked on an equal footing as others

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Lung-healthy group: 5 persons will be recruited via bulletins in staff rooms and outpatient clinics at participating departments/hospitals.
  Bronchiectasis group: 5 patients will be recruited via outpatient clinics at participating departments/hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Changes in air temperature | 1 day
  Changes in air temperature (under 88-92℃ surroundings) measured in both lungs at 1st, 2nd and 3rd bronchial segment, at 4th and 5th bronchial segment and at 6th-10th. bronchial segment at times 0 s, 15 s, 30 s, 45 s, 60 s, 75 s, 90 s, 105 s, 120 s, 135 s, and 150 s.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine, Section of Respiratory Medicine, Herlev and Gentofte Hospital, Gentofte Municipality, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP